CLINICAL TRIAL: NCT05400993
Title: A Multicenter, Single-arm Prospective Phase II Study of Chidamide in Combination With Chemotherapy for Neoadjuvant Treatment of HR-positive/HER2-negative Breast Cancer
Brief Title: Clinical Study of Chidamide Combined With Chemotherapy in Neoadjuvant Treatment of HR+/ HER2-BC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Postdoctoral 、chief physician, Shengjing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-C25
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Epirubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Chidamide combined with EC -- T regimen was treated with 1 cycle every 21 days, followed by 4 cycles of EC followed by 4 cycles of T, a total of 8 cycles
  Interventions: Combination Product: Chidamide

INTERVENTIONS:
Combination Product: Chidamide — Chidamide: take orally twice a week,4 tablets/time (20mg/ time), the interval between two doses should not be less than 3 days (such as Monday and Thursday, Tuesday and Friday, Wednesday and Saturday, etc.), the day before chemotherapy, 30 minutes after breakfast； Chidamide: 20mg, orally, twice a week, oral for two weeks and one week, a total of 8 cycles； Epirubicin 90mg/m2 , ivgtt, d1 Cyclophosphamide 600mg/m 2, ivgtt, d1 Q3w, 4 cycle； sequential Docetaxel 100 mg/m 2, IVGtt, D1 Q3w, 4 cycle。
  Other Names: pharmorubicin; Cyclophosphamide; Docetaxel

SUMMARY:
Neoadjuvant therapy for HR+/HER2- breast cancer is dominated by anthracycline combined with paclitaxel chemotherapy. Aggressive neoadjuvant chemotherapy can only achieve pCR in about 10% of PATIENTS with HR-positive breast cancer. The emergence of new targeted drugs brings new life and hope to HR-positive breast cancer patients.Basic studies have shown that the abnormal state of epigenetics is associated with the metastasis of drug resistance and recurrence of tumor histone deacetylase (HDAC) is an important regulator of epigenetic regulation, and drugs targeting HDAC provide a new strategy for tumor therapy. The ACE study suggests that selective HDAC inhibitor chidamide in combination with endocrine therapy significantly improves survival benefit in patients with hr-positive HER2-negative advanced breast cancer who relapsed or progressed after endocrine therapy, providing a new treatment option for these patients.In conclusion, we hypothesize that neoadjuvant therapy with chidamide combination therapy provides a better strategy for patients with HR + /HER2 - breast adenocarcinoma.

DETAILED DESCRIPTION:
A total of 59 patients with stage Ii-III HR + / HER2 - breast cancer were enrolled in a multi-center, single-arm prospective design. The main purpose of the study was to observe the efficacy and safety of chidamide combined with chemotherapy in neoadjuvant treatment of stage II-III HR + / HER2 - breast cancer Breast MRI and other imaging examinations were reviewed every 2 cycles to evaluate the efficacy. If the efficacy was accurate, surgical treatment was performed within 4 weeks after the 8th cycle of neoadjuvant therapy. If the efficacy was SD+/PD, the study would be withdrawn Within 4 weeks after surgical treatment, the resected tumor tissue and lymph nodes were histopathologically examined (including the pathology of the tumor resection margin). The pathological sections were uniformly lent to the master research unit for unified review

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years or older and 75 years or younger;
2. All patients were histopathologically confirmed to be estrogen receptor (ER) positive (& GT; 10%),HER2 receptor negative follows the 2018 ASCO-CAP HER2 negative interpretation guideline criteria;
3. Newly treated patients with stage II-III tumor staging meeting AJCC Version 8 criteria;
4. KPS score ≥70;
5. The functional level of the organ must meet the following requirements:

   * Bone marrow function
   * ANC ≥ 1.5×10 9 /L (growth factor not used within 14 days);
   * PLT ≥ 100×10 9 /L (no corrective treatment within 7 days);
   * Hb ≥ 100 g/L (no corrective treatment within 7 days);
   * Liver and kidney function
   * TBIL ≤1.5 x ULN;
   * ALT and AST≤3×ULN;
   * BUN and Cr≤1.5×ULN and creatinine clearance ≥50 mL/min (Cockcroft-Gault formula);
6. Able to undergo needle biopsy;
7. Volunteered to participate in the study, signed informed consent, had good compliance and was willing to cooperate with follow-up.

Exclusion Criteria:

-

Participants are not allowed to participate in the clinical study under any of the following conditions:

1. Have received any other form of anti-tumor therapy (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.);
2. Receiving any other antitumor therapy;
3. Bilateral breast cancer, inflammatory breast cancer or ocessive breast cancer;
4. Stage IV breast cancer;
5. Breast cancer without histopathological diagnosis;
6. Other malignant tumors within the past 5 years, except cured carcinoma in situ of the cervix;
7. Severe heart, liver, kidney and other important organ dysfunction;
8. Inability to swallow, chronic diarrhea and intestinal obstruction, there are many factors affecting drug taking and absorption;
9. Participated in clinical trials of other drugs within 4 weeks before enrollment;
10. Known history of allergy to the drug components of this regimen; History of immunodeficiency, including HIV positive, HCV, live active hepatitis B or other acquired or congenital immune deficiency diseases, or a history of organ transplantation;
11. History of any heart disease, including :(1) medically required or clinically significant arrhythmia; (2) myocardium infarction; (3) heart failure; (4) Any other heart disease deemed unsuitable for the study by the investigator;
12. Pregnant, lactating women, fertile women with positive baseline pregnancy test or in the entire women of reproductive age who were unwilling to use effective contraception during the trial;
13. According to the investigator's judgment, there are comorbidities (including but) that seriously endanger the patient's safety or affect the patient's ability to complete the study not limited to severe hypertension, severe diabetes, active infection, etc., which cannot be controlled by drugs);
14. A clear past history of neurological or psychiatric disorders, including epilepsy or dementia. The investigator considered the patient unsuitable for the study in any other case.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-05-23 (Estimated); Study Completion 2024-05-23 (Estimated)

PRIMARY OUTCOMES:
RCB 0-1 points ratio | One month after surgery
  Residual tumor burden

SECONDARY OUTCOMES:
pCR（ypT0/is、ypN0） | One month after surgery
  There was no residual tumor
bpCR（ypT0/is） | One month after surgery
  Breast pCRwith ypT0/is carcinoma in situ
ORR | Period of neoadjuvant therapy (treatment 1-6 months)
  Proportion of patients who had a 30% reduction in tumor volume and maintained it for more than four weeks
Breast retention rate | One month after surgery
  Percentage of patients with successful breast preservation

OTHER OUTCOMES:
Adverse Events (AE) and Serious Adverse Events (SAE) | Period of neoadjuvant therapy (treatment 1-6 months)And chidamide 3 weeks after withdrawal
  Any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, doctoral, Principal Investigator — Shengjing Hospital
Locations (7):
- China (7):
  - Cancer Hospital affiliated to Harbin Medical University, Haerbin, Heilongjiang
  - Bethune First Hospital of Jilin University, Changchun, Jilin
  - Health Science and Technology Information Center of Liaoning Health Industry Group Co., LTD, Benxi, Liaoning
  - Affiliated Zhongshan Hospital Dalian University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning

REFERENCES:
- [Derived] Xue J, Shan H, Qiu F, Niu N, Chen G, Xu Q, Gu X, Xing F, Xu Y, Zheng X, He G, Xu H, Zhang H, Song D, Han Y, Tang M, Cao S, Song Y, Zheng R, Zhao Y, Jiao G, Liu M, Liu C. Neoadjuvant chidamide combined with chemotherapy in patients with hormone receptor-positive, human epidermal growth factor receptor 2-negative breast cancer (MUKDEN 05): a multicentre, single-arm, phase 2 trial. Lancet Reg Health West Pac. 2025 Sep 27;63:101700. doi: 10.1016/j.lanwpc.2025.101700. eCollection 2025 Oct. PMID 41080407